CLINICAL TRIAL: NCT06744634
Title: An Analysis of Factors Associated with Chronic Musculoskeletal Pain, Pain Management Preferences, Coping Strategies and Health-related Quality of Life Among Older People: a Comparative Cross-Cultural Study of Turkey, Croatia and Romania
Brief Title: Coping Strategies with Pain Among Older People
Acronym: Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Assis. Dr., Biruni University
Other Study IDs: Coping strategies; Biruni U (Registry Identifier: Coping strategies with pain)
Record Dates: First submitted 2024-12-11; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pain
Keywords: Aged; Coping Strategy; Health-Related Quality of Life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Romania Group: The structured questionnaire was performed by older adults from Romania
  Interventions: Other: Romania group
- Turkey Group: The structured questionnaire was performed by older adults from Turkey
  Interventions: Other: Turkey Group
- Croatia Group: The structured questionnaire was performed by older adults from Croatia
  Interventions: Other: Croatia Group

INTERVENTIONS:
Other: Romania group — The questionnaire which was prepared by researchers will be performed by older adults from Romania. The sociodemographic characteristics are recorded to part A section of questionnaire. The pain assessment section is part B and evaluate pain localization, intensity, type, factors affecting the pain, coping and management strategies of pain. Health related outcomes will be evaluated with CDC (Center of Disease Control and Prevention) Health related Quality of Life-4 Questionnaire
  Groups: Romania Group
Other: Turkey Group — The questionnaire which was prepared by researchers will be performed by older adults from Turkey The sociodemographic characteristics are recorded to part A section of questionnaire. The pain assessment section is part B and evaluate pain localization, intensity, type, factors affecting the pain, coping and management strategies of pain. Health related outcomes will be evaluated with CDC (Center of Disease Control and Prevention) Health related Quality of Life-4 Questionnaire
  Groups: Turkey Group
Other: Croatia Group — The questionnaire which was prepared by researchers will be performed by older adults from Croatia. The sociodemographic characteristics are recorded to part A section of questionnaire. The pain assessment section is part B and evaluate pain localization, intensity, type, factors affecting the pain, coping and management strategies of pain. Health related outcomes will be evaluated with CDC (Center of Disease Control and Prevention) Health related Quality of Life-4 Questionnaire
  Groups: Croatia Group

SUMMARY:
Chronic musculoskeletal pain is common among older adults. This study aimed to identify and describe the characteristics of chronic musculoskeletal pain, pain management and coping strategies among older adults from Turkey, Croatia and Romania. The study also aimed to explore cultural differences in pain experience and management.

Methods:

337 older adults with chronic pain participate 100 from Turkey, 131 from Croatia and 106 from Romania. Semi-structured interviews will explore four main topics, including factors influencing pain, coping strategies, management strategies, and health-related quality of life.

DETAILED DESCRIPTION:
The questionnaire which was prepared by researchers will be performed by older adults. The sociodemographic characteristics are recorded to part A section of questionnaire. The pain assessment section is part B and evaluate pain localization, intensity, type, factors affecting the pain, coping and management strategies of pain. Health related outcomes will be evaluated with CDC (Center of Disease Control and Prevention) Health related Quality of Life-4 Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* women and men aged between 65-85 years
* living in their own homes or in a nursing home
* older adults with chronic pain for at least 6 months,
* independent in activities of daily living, and independent in walking (with or without assistive walking devices).

Exclusion Criteria:

* Elderly adults with communication problems

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Geriatrics
Sampling Method: Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
A semi-structure questionnaire | 1 week
  Four main themes were
  identified: (i) the factors affecting pain such as increasing and decreasing factors in ageing; (ii) the coping strategies with pain in ageing; (iii) the management strategies in ageing; (iv) the health related quality of life related pain in ageing
Visuel analog scale | 1 week
  The VAS is a tool for measuring subjective experiences like pain, discomfort, or other sensations, commonly used with older adults in clinical settings. It helps assess pain intensity, especially in those with communication challenges due to cognitive decline or sensory impairment. VAS is useful for evaluating pain severity in conditions like osteoarthritis, neuropathy, post-surgical pain, and cancer-related pain In this study, participants will rate their pain on an 11-point scale, from 0 (no pain) to 10 (worst pain imaginable). Scores were categorized as severe (7-10), moderate (4-6,9), mild (1-3,9), or no pain (0)

SECONDARY OUTCOMES:
CDC Health related Quality of Life-4 | 1 week
  develop to assess a person s sense of well-being through four questions. A core set of these measures (the CDC HRQOL-4) asks about self-rated general health and the number of recent days when a person is physically unhealthy, mentally unhealthy, or limited in usual activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Istanbul, Turkey (Türkiye)